CLINICAL TRIAL: NCT02111343
Title: Pilot Study: The Effectiveness of Computerized Auditory Training Programme on Children With Auditory Processing Disorder
Brief Title: The Effectiveness of Computerized Auditory Training Programme on Children With Auditory Processing Disorder
Acronym: CBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Dr. Jenny Loo, Principal Audiologist, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D/09/485
Record Dates: First submitted 2014-03-25; First posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Central Auditory Processing Disorder
Keywords: auditory processing disorder; central auditory processing disorder; auditory processing; auditory training
MeSH Terms: conditions — Language Development Disorders; Auditory Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer-based auditory training (CBAT) (Experimental): The CBAT programmes in the current study were specifically designed to improve speech-in-noise and dichotic listening skills of children diagnosed with CAPD. All the training programmes were designed to be installed on home-user's computer, and they were visually attractive and appealing to children. The development of the software (non commercial) for the speech-in-noise and dichotic listening training was done by two different teams in the United Kingdom and Singapore, respectively.
  Interventions: Other: Computer-based auditory training (CBAT)
- Control (No Intervention): No intervention other than participants' regular school activities

INTERVENTIONS:
Other: Computer-based auditory training (CBAT) — There are 3 listening games (i.e. Doggy, Who-Is-Right, Story-in-noise) that target on speech-in-noise training and 1 listening game (i.e. TATP) that aims to train dichotic listening.
  Patient was required to undergo the training for 30 minutes per day, 5 sessions per week, for a duration of 12 weeks. Parents were advised to keep a journal to record child's training hour of the day.
  Arms: Computer-based auditory training (CBAT)

SUMMARY:
The current study aimed to examine the effectiveness of a Computer-based auditory training (CBAT) intervention for children with Central Auditory Processing Disorder (CAPD) by comparing the changes in auditory processing (AP) and functional listening skills of these children immediately post-intervention, to that of the untrained controls. The AP skills of the trained group were evaluated again at 3 months post-intervention to examine the sustainability of any improvements made from the CBAT intervention. I hypothesised that after intervention, children from the auditory training (AT) group would improve in their AP skills, and that improvement would be greater than the changes in AP skills of those untrained controls. I also hypothesised that the improvement made from the intervention would sustain for at least 3 months after the end of intervention. Finally, I examined if the training outcomes are predictable from any underlying factors such as the initial AP, language, or cognitive skills of these children.

DETAILED DESCRIPTION:
This prospective study incorporated a parallel group design that randomly assigned participants identified with CAPD to an auditory training (AT) group or a no intervention (Control) group. Both groups were matched for age and gender. Baseline measures were conducted prior to the randomisation process.

Participants from the AT group were given a 3-month home therapy using a CBAT programme developed for this study, while participants from the control group received no intervention for the same period of time. Apart from regular school attendance and activities, all participants were requested to discontinue any other auditory-based interventions, which might affect the outcomes of this study. All the participants were assessed again after the conclusion of the training period.

After the end of the intervention, participants from the AT group were requested to undergo a no-intervention phase for a period of 3 months before another assessment. This was intended to examine the sustainability of any improvement made through the CBAT programme.

An auditory test and two validated questionnaires were used as outcome measures, administered at baseline, and at post-3 months (immediately post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Presentation to the clinic with reported symptoms of listening difficulties.
* No measurable peripheral hearing anomalies in both ears, i.e. normal cochlea and middle ear function, as judged by normal audiometric thresholds of 20dB HL or better in the speech frequency range of 250-8000 Hz, and normal impedance audiometry.
* Performance on the behavioural AP test battery (Table 6.1) which met the following criteria:

  * At least two abnormalities in the non-speech or minimally-linguistic loaded tasks.
  * No indication of any other underlying higher order cognitive problems as judged by abnormal performance scores in all the tasks in AP test battery.
* Normal intelligence, as judged by having a nonverbal IQ score of more than 85 (Test of Nonverbal Intelligence, TONI).

Exclusion Criteria:

* one with medical or developmental conditions, i.e. epilepsy, global developmental delay, pervasive learning disorder such as autism, which may additionally impact on auditory or cognitive performance.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in auditory processing skills at 3 months | baseline, and post-3 months
  The auditory processing skills of patients were assessed using the LiSN-S. The LiSN-S is an auditory task that assesses the ability of children to understand speech in the background of two other talkers. The LiSN-S test was administered using a laptop with a circumaural headphones connected to the computer. The target sentences were presented at an initial level of 62 dB SPL, whereas the distracter stories were presented at a constant level of 55 dB SPL. The target stimuli and distracter discourse were presented to both ears simultaneously. A maximum of 30 sentences were presented in each of the four listening conditions. The patient was required to repeat the targeted sentences verbally in every listening condition and correct responses were scored manually by the me on the computer. The stimulus presentation level was adjusted adaptively depending on the patient's response. The assessment took approximately 20 minutes to complete.

SECONDARY OUTCOMES:
Change from baseline in listening skills at 3 months | Baseline, and post-3 months
  The listening skills of patients were assessed using two questionnaires: a) Pragmatic Profile (PP) questionnaire consisted of 52 items concerning the rituals and conversational skills of a child, how a child asks for information and gives responses, and nonverbal communication skills; b) The CHAPS questionnaire consisted of 36 questions evaluating a child's listening skills in 6 different auditory conditions (noise, quiet, ideal, multiple inputs, auditory memory sequencing, and auditory attention span) in comparison to his/her peers. The PP and CHAPS questionnaire was completed by each patient's parents and teacher respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny HY Loo, PhD, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore